CLINICAL TRIAL: NCT01775527
Title: IgA Nephropathy, Lymphocyte Homing and IgA Class Switch
Acronym: NIDOCIGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: I10 014
Record Dates: First submitted 2013-01-18; First posted 2013-01-25 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2012-11

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- blood test (Other)
  Interventions: Other: blood test

INTERVENTIONS:
Other: blood test

SUMMARY:
IgA nephropathy (IgAN) is the most common primary glomerulonephritis in the world and it represents an important cause of end-stage kidney failure. This disease was described as a distinct entity in 1968 by J Berger and N Hinglais. The aetiology and the pathogenesis remain still obscure. Clinical observations and immunisation studies indicate that IgAN represents a dysregulation of the immune system, rather than an intrinsic renal abnormality. Twenty years ago, some authors proposed the mucosa-bone marrow axis to explain the pathogenesis of the disease. Mucosal IgA plasmocytes are displaced and take up residence in systemic sites. The unusual characteristics featured by the IgA produced by these cells (charge, size, glycosylation) drive their accumulation, deposition and mesangial activation characteristic of IgAN.

Evidence is emerging that altered lymphocyte homing may ultimately explain this aberrant localization.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 70 years
* IgA nephropathy documented by the kidney biopsy in the six months preceding the inclusion
* Glomerular filtration rate (MDRD formula as simplified) < 90 ml/mn and > 30 ml/mn/1,73 m2
* Consent form signed

Exclusion Criteria:

* Patients with cirrhosis or chronic liver disease
* Patients with a history of Crohn's disease or celiac disease
* Patients who received treatment with corticosteroids or affiliates for six months
* Patients who received a live attenuated vaccine during the past 4 weeks
* Patients with a known infection such as HIV, hepatitis B or C
* Patients who presented with a serious infection during the last month
* Breastfeeding women
* Patients not affiliated with a social security scheme
* Under guardianship patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Primary Outcome Measure of this study is the level of expression of the molecules of intestinal localization. | 30 minutes

SECONDARY OUTCOMES:
The secondary outcome measure is the level of expression of the homing molecules in lymphocytes B IgA memory | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Boumediene, doctor, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, Limoges, France